CLINICAL TRIAL: NCT03981029
Title: Folic Acid Clinical Trial (FACT): Biomarker Subgroup Analysis
Brief Title: FACT Biomarker Subgroup Analysis
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2011649-01H
Record Dates: First submitted 2019-06-03; First posted 2019-06-10 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2019-06

CONDITIONS: Pre-Eclampsia
Keywords: Folate; One Carbon Metabolism; Preeclampsia; Folic Acid; Pregnancy
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral Whole Blood, Plasma, Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FACT High-dose folic acid treatment group: Consenting study participants who, through their participation in FACT (NCT01355159) are randomized to receive daily high-dose folic acid supplementation during pregnancy.
  Interventions: Other: 4.0mg Folic Acid received through participation in FACT (NCT01355159)
- FACT Placebo treatment group: Consenting study participants who, through their participation in FACT (NCT01355159) are randomized to receive daily placebo supplementation during pregnancy.
  Interventions: Other: Placebo received through participation in FACT

INTERVENTIONS:
Other: 4.0mg Folic Acid received through participation in FACT (NCT01355159) — Participants in this study received either daily high-dose folic acid supplementation during pregnancy OR placebo through their participation in FACT (NCT01355159). Details of the FACT Folic Acid intervention are provided below:
  Folic Acid 1.0 mg x 4 tablets will be taken daily by oral administration. The majority of women in the study will routinely take 1.0 mg folic acid in a prenatal vitamin supplement, as recommended by their primary obstetrical provider; the study requirements do not require that participants change their practice. Therefore the actual total daily dose may be up to 5.1 mg of folic acid
  Groups: FACT High-dose folic acid treatment group
Other: Placebo received through participation in FACT — Participants in this study received either daily high-dose folic acid supplementation during pregnancy OR placebo through their participation in FACT (NCT01355159). Details of the FACT Folic Acid placebo are provided below:
  Placebo x 4 tablets will be taken daily by oral administration.
  Groups: FACT Placebo treatment group

SUMMARY:
The FACT Biomarker Subgroup Analysis is a pilot study of mothers who participated in the Folic Acid Clinical Trial (FACT, NCT01355159). This subgroup analysis aims to determine the effect of high-dose folic acid supplementation in pregnancy on maternal folate status and subsequent impact on risk for pre-eclampsia.

DETAILED DESCRIPTION:
The Folic Acid Clinical Trial (FACT) was developed to conclusively determine the effect of high dose folic acid supplementation in pregnancy on the prevention of preeclampsia (PE) in a randomized controlled trial (RCT) design.

The primary objective of the FACT Biomarker Subgroup Analysis is to determine the folate status and its impact on risk for PE in a subgroup of women participating in FACT. Our secondary objectives are to:

i) To determine serum vitamin B6 and B12 status, modifiers of folate metabolism, and their impact on risk for PE in women participating in the FACT

ii) To determine plasma homocysteine status, a folate-responsive biomarker for PE risk, and its relationship with risk for PE in women participating in the FACT

iii) To determine the modifying effect of single nucleotide polymorphisms (SNPs) in key folate metabolic enzymes (MTHFR, MTHFD1, MTR) on PE risk in women participating in the FACT

iv) To determine the effect of folic acid supplementation and folate status on biomarkers of PE (sFLT, sENG, PlGF) and their association with PE risk in women participating in the FACT

Folate biomarker analyses will provide key information to identify modifiers of the response to folic acid treatment and elucidate the mechanism(s) underlying the relationship between folic acid treatment and PE risk. Folate status will vary in response to folic acid treatment depending on a number of factors including compliance in taking the study supplement, folate intake from the diet (natural folate and folic acid used for enrichment), vitamin B12 status, and genetic polymorphisms in enzymes involved in folate metabolism that have been shown to effect placental development/function. As such, variation in the response to folic acid treatment may account for differences in observed PE risk.

Folic acid supplementation may also reduce homocysteine, its related endothelial dysfunction and consequently reduce PE risk. In addition, homocysteine metabolism is dependent on vitamins B12 and B6, the deficiency of which can result in hyperhomocysteinemia. Thus, homocysteine, B12 and B6 will each be evaluated.

Lastly, it will be useful to assess biomarkers of placental health and PE risk (sFlt-1, sEng, PlGF) that are found in maternal circulation and determine their association with folate intake and status.

ELIGIBILITY:
Individuals participating in FACT (NCT01355159) will be eligible to participate. FACT eligibility criteria are as follows:

INCLUSION criteria

1. Capability of subject to comprehend and comply with study requirements
2. ≥ 18 years of age at time of consent
3. Subject is taking ≤1.1 mg of folic acid daily at the time of randomization
4. Live fetus (documented positive fetal heart prior to randomization)
5. Gestational age between 8+0 and 16+6 weeks of pregnancy (Gestational age (GA) of subjects will be calculated based on the first day of the last menstrual period (LMP) or ultrasound performed before 12+6. If early ultrasound and LMP dates differ by ≤ 7 days, base GA estimate on LMP date; if > 7 days, use early < 12+6 ultrasound)
6. Subject plans to give birth in a participating hospital site
7. Pregnant subjects must fulfill at least one of the following identified risk factors for pre-eclampsia (PE):

   * Pre-existing hypertension (documented evidence of diastolic blood pressure ≥ 90 mmHg on two separate occasions or at least 4 hours apart prior to randomization, or use of antihypertensive medication during this pregnancy specifically for the treatment of hypertension prior to randomization)
   * Pre-pregnancy diabetes (documented evidence of Type I or type II DM)
   * Twin pregnancy
   * Documented evidence of history of PE in a previous pregnancy
   * BMI > 35 kg/m2 within 3 months prior to this pregnancy and up to randomization of this pregnancy (documented evidence of height and weight to calculate BMI is required)

EXCLUSION Criteria:

1. Known history or presence of any clinically significant disease or condition which would be a contraindication to folic acid supplementation of up to 5 mg daily for the duration of pregnancy
2. Known major fetal anomaly or fetal demise
3. History of medical complications, including: renal disease with altered renal function, epilepsy, cancer, or use of folic acid antagonists such as valproic acid
4. Individual who is currently enrolled or has participated in another clinical trial or who received an investigational drug within 3 months of the date of randomization (unless approved by the Trial Coordinating Centre)
5. Known presence of: Alcohol abuse (≥ 2 drinks per day) or alcohol dependence, Illicit drug/substance use and/or dependence, Known hypersensitivity to folic acid, Multiple Pregnancy (triplets or more), Participation in this study in a previous pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The FACT Biomarker Subgroup Analysis is a pilot study that aims to determine the folate status and its impact on risk for pre-eclampsia in a subgroup of women participating in FACT (NCT01355159).
  Women participating in FACT (NCT01355159) will be eligible to participate.
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2011-12-19 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - The Moncton Hospital, Moncton, New Brunswick
  - Kingston General Hospital, Kingston, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Health Canada, Ottawa, Ontario

REFERENCES:
- [Background] Wen SW, White RR, Rybak N, Gaudet LM, Robson S, Hague W, Simms-Stewart D, Carroli G, Smith G, Fraser WD, Wells G, Davidge ST, Kingdom J, Coyle D, Fergusson D, Corsi DJ, Champagne J, Sabri E, Ramsay T, Mol BWJ, Oudijk MA, Walker MC; FACT Collaborating Group. Effect of high dose folic acid supplementation in pregnancy on pre-eclampsia (FACT): double blind, phase III, randomised controlled, international, multicentre trial. BMJ. 2018 Sep 12;362:k3478. doi: 10.1136/bmj.k3478. PMID 30209050
- [Background] Wen SW, Chen XK, Rodger M, White RR, Yang Q, Smith GN, Sigal RJ, Perkins SL, Walker MC. Folic acid supplementation in early second trimester and the risk of preeclampsia. Am J Obstet Gynecol. 2008 Jan;198(1):45.e1-7. doi: 10.1016/j.ajog.2007.06.067. PMID 18166303
- [Background] Shane B, Stokstad EL. Vitamin B12-folate interrelationships. Annu Rev Nutr. 1985;5:115-41. doi: 10.1146/annurev.nu.05.070185.000555. PMID 3927946
- [Background] Guven MA, Coskun A, Ertas IE, Aral M, Zencirci B, Oksuz H. Association of maternal serum CRP, IL-6, TNF-alpha, homocysteine, folic acid and vitamin B12 levels with the severity of preeclampsia and fetal birth weight. Hypertens Pregnancy. 2009 May;28(2):190-200. doi: 10.1080/10641950802601179. PMID 19437229
- [Background] Lindblad B, Zaman S, Malik A, Martin H, Ekstrom AM, Amu S, Holmgren A, Norman M. Folate, vitamin B12, and homocysteine levels in South Asian women with growth-retarded fetuses. Acta Obstet Gynecol Scand. 2005 Nov;84(11):1055-61. doi: 10.1111/j.0001-6349.2005.00876.x. PMID 16232172
- [Background] Dalery K, Lussier-Cacan S, Selhub J, Davignon J, Latour Y, Genest J Jr. Homocysteine and coronary artery disease in French Canadian subjects: relation with vitamins B12, B6, pyridoxal phosphate, and folate. Am J Cardiol. 1995 Jun 1;75(16):1107-11. doi: 10.1016/s0002-9149(99)80739-5. PMID 7762494
- [Background] Powers RW, Evans RW, Majors AK, Ojimba JI, Ness RB, Crombleholme WR, Roberts JM. Plasma homocysteine concentration is increased in preeclampsia and is associated with evidence of endothelial activation. Am J Obstet Gynecol. 1998 Dec;179(6 Pt 1):1605-11. doi: 10.1016/s0002-9378(98)70033-x. PMID 9855605
- [Background] Stover PJ. Physiology of folate and vitamin B12 in health and disease. Nutr Rev. 2004 Jun;62(6 Pt 2):S3-12; discussion S13. doi: 10.1111/j.1753-4887.2004.tb00070.x. PMID 15298442
- [Background] Hustad S, Midttun O, Schneede J, Vollset SE, Grotmol T, Ueland PM. The methylenetetrahydrofolate reductase 677C-->T polymorphism as a modulator of a B vitamin network with major effects on homocysteine metabolism. Am J Hum Genet. 2007 May;80(5):846-55. doi: 10.1086/513520. Epub 2007 Mar 13. PMID 17436239
- [Background] Parle-McDermott A, Kirke PN, Mills JL, Molloy AM, Cox C, O'Leary VB, Pangilinan F, Conley M, Cleary L, Brody LC, Scott JM. Confirmation of the R653Q polymorphism of the trifunctional C1-synthase enzyme as a maternal risk for neural tube defects in the Irish population. Eur J Hum Genet. 2006 Jun;14(6):768-72. doi: 10.1038/sj.ejhg.5201603. PMID 16552426
- [Background] Parle-McDermott A, Mills JL, Kirke PN, Cox C, Signore CC, Kirke S, Molloy AM, O'Leary VB, Pangilinan FJ, O'Herlihy C, Brody LC, Scott JM. MTHFD1 R653Q polymorphism is a maternal genetic risk factor for severe abruptio placentae. Am J Med Genet A. 2005 Feb 1;132A(4):365-8. doi: 10.1002/ajmg.a.30354. PMID 15633187
- [Background] Parle-McDermott A, Pangilinan F, Mills JL, Signore CC, Molloy AM, Cotter A, Conley M, Cox C, Kirke PN, Scott JM, Brody LC. A polymorphism in the MTHFD1 gene increases a mother's risk of having an unexplained second trimester pregnancy loss. Mol Hum Reprod. 2005 Jul;11(7):477-80. doi: 10.1093/molehr/gah204. PMID 16123074
- [Background] Furness DL, Fenech MF, Khong YT, Romero R, Dekker GA. One-carbon metabolism enzyme polymorphisms and uteroplacental insufficiency. Am J Obstet Gynecol. 2008 Sep;199(3):276.e1-8. doi: 10.1016/j.ajog.2008.06.020. PMID 18771981
- [Background] Tam LE, McDonald SD, Wen SW, Smith GN, Windrim RC, Walker MC. A survey of preconceptional folic acid use in a group of Canadian women. J Obstet Gynaecol Can. 2005 Mar;27(3):232-6. doi: 10.1016/s1701-2163(16)30515-1. PMID 15937596
- [Background] Shakur YA, Garriguet D, Corey P, O'Connor DL. Folic acid fortification above mandated levels results in a low prevalence of folate inadequacy among Canadians. Am J Clin Nutr. 2010 Oct;92(4):818-25. doi: 10.3945/ajcn.2010.29696. Epub 2010 Aug 25. PMID 20739423
- [Background] Czeizel AE, Tomcsik M. Acute toxicity of folic acid in pregnant women. Teratology. 1999 Jul;60(1):3-4. doi: 10.1002/(SICI)1096-9926(199907)60:13.0.CO;2-4. No abstract available. PMID 10413330
- [Background] Czeizel AE, Dudas I, Metneki J. Pregnancy outcomes in a randomised controlled trial of periconceptional multivitamin supplementation. Final report. Arch Gynecol Obstet. 1994;255(3):131-9. doi: 10.1007/BF02390940. PMID 7979565
- [Background] Czeizel AE, Susanszky E. Diet intake and vitamin supplement use of Hungarian women during the preconceptional period. Int J Vitam Nutr Res. 1994;64(4):300-5. PMID 7883469
- [Background] Ericson A, Kallen B, Aberg A. Use of multivitamins and folic acid in early pregnancy and multiple births in Sweden. Twin Res. 2001 Apr;4(2):63-6. doi: 10.1375/1369052012155. PMID 11665336
- [Background] Kirke PN, Daly LE, Elwood JH. A randomised trial of low dose folic acid to prevent neural tube defects. The Irish Vitamin Study Group. Arch Dis Child. 1992 Dec;67(12):1442-6. doi: 10.1136/adc.67.12.1442. PMID 1489222
- [Background] Stevens VL, McCullough ML, Sun J, Gapstur SM. Folate and other one-carbon metabolism-related nutrients and risk of postmenopausal breast cancer in the Cancer Prevention Study II Nutrition Cohort. Am J Clin Nutr. 2010 Jun;91(6):1708-15. doi: 10.3945/ajcn.2009.28553. Epub 2010 Apr 21. PMID 20410093
- [Background] Wu K, Helzlsouer KJ, Comstock GW, Hoffman SC, Nadeau MR, Selhub J. A prospective study on folate, B12, and pyridoxal 5'-phosphate (B6) and breast cancer. Cancer Epidemiol Biomarkers Prev. 1999 Mar;8(3):209-17. PMID 10090298
- [Background] Zhang SM, Cook NR, Albert CM, Gaziano JM, Buring JE, Manson JE. Effect of combined folic acid, vitamin B6, and vitamin B12 on cancer risk in women: a randomized trial. JAMA. 2008 Nov 5;300(17):2012-21. doi: 10.1001/jama.2008.555. PMID 18984888
- [Background] Zhang SM, Willett WC, Selhub J, Hunter DJ, Giovannucci EL, Holmes MD, Colditz GA, Hankinson SE. Plasma folate, vitamin B6, vitamin B12, homocysteine, and risk of breast cancer. J Natl Cancer Inst. 2003 Mar 5;95(5):373-80. doi: 10.1093/jnci/95.5.373. PMID 12618502
- [Background] Larsson SC, Giovannucci E, Wolk A. Folate and risk of breast cancer: a meta-analysis. J Natl Cancer Inst. 2007 Jan 3;99(1):64-76. doi: 10.1093/jnci/djk006. PMID 17202114
- [Background] Figueiredo JC, Mott LA, Giovannucci E, Wu K, Cole B, Grainge MJ, Logan RF, Baron JA. Folic acid and prevention of colorectal adenomas: a combined analysis of randomized clinical trials. Int J Cancer. 2011 Jul 1;129(1):192-203. doi: 10.1002/ijc.25872. Epub 2011 Apr 1. PMID 21170989
- [Background] Kim DH, Smith-Warner SA, Spiegelman D, Yaun SS, Colditz GA, Freudenheim JL, Giovannucci E, Goldbohm RA, Graham S, Harnack L, Jacobs EJ, Leitzmann M, Mannisto S, Miller AB, Potter JD, Rohan TE, Schatzkin A, Speizer FE, Stevens VL, Stolzenberg-Solomon R, Terry P, Toniolo P, Weijenberg MP, Willett WC, Wolk A, Zeleniuch-Jacquotte A, Hunter DJ. Pooled analyses of 13 prospective cohort studies on folate intake and colon cancer. Cancer Causes Control. 2010 Nov;21(11):1919-30. doi: 10.1007/s10552-010-9620-8. Epub 2010 Sep 5. PMID 20820900
- [Background] Mills JL, Von Kohorn I, Conley MR, Zeller JA, Cox C, Williamson RE, Dufour DR. Low vitamin B-12 concentrations in patients without anemia: the effect of folic acid fortification of grain. Am J Clin Nutr. 2003 Jun;77(6):1474-7. doi: 10.1093/ajcn/77.6.1474. PMID 12791626
- [Background] Wilson RD; GENETICS COMMITTEE; MOTHERISK. RETIRED: Pre-conceptional vitamin/folic acid supplementation 2007: the use of folic acid in combination with a multivitamin supplement for the prevention of neural tube defects and other congenital anomalies. J Obstet Gynaecol Can. 2007 Dec;29(12):1003-1013. doi: 10.1016/S1701-2163(16)32685-8. English, French. PMID 18053387
- See also: High Dose Folic Acid Supplementation Throughout Pregnancy for Preeclampsia Prevention (FACT) ClinicalTrials.gov registration — https://clinicaltrials.gov/ct2/show/NCT01355159

RESULTS

PARTICIPANT FLOW:
Groups:
- FACT High-dose Folic Acid Treatment Group: Consenting study participants who, through their participation in FACT (NCT01355159) are randomized to receive daily high-dose folic acid supplementation during pregnancy.
  4.0mg Folic Acid received through participation in FACT (NCT01355159): Participants in this study received either daily high-dose folic acid supplementation during pregnancy OR placebo through their participation in FACT (NCT01355159). Details of the FACT Folic Acid intervention are provided below:
  Folic Acid 1.0 mg x 4 tablets will be taken daily by oral administration. The majority of women in the study will routinely take 1.0 mg folic acid in a prenatal vitamin supplement, as recommended by their primary obstetrical provider; the study requirements do not require that participants change their practice. Therefore the actual total daily dose may be up to 5.1 mg of folic acid
- FACT Placebo Treatment Group: Consenting study participants who, through their participation in FACT (NCT01355159) are randomized to receive daily placebo supplementation during pregnancy.
  Placebo received through participation in FACT: Participants in this study received either daily high-dose folic acid supplementation during pregnancy OR placebo through their participation in FACT (NCT01355159). Details of the FACT Folic Acid placebo are provided below:
  Placebo x 4 tablets will be taken daily by oral administration.
Period: Overall Study
Arm/Group | FACT High-dose Folic Acid Treatment Group | FACT Placebo Treatment Group
Started | 19 | 32
Completed | 19 | 31
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FACT High-dose Folic Acid Treatment Group | FACT Placebo Treatment Group | Total
Number analyzed (Participants) | 19 | 31 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [30 to 37] | 32 [28 to 34] | 32 [30 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 31 | 50
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian race | 18 | 28 | 46
  Other race | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 19 | 31 | 50

OUTCOME MEASURES:

1. Primary Outcome: Folate Status
Description: The primary outcome measure is maternal folate status. Folate status will be determined by:
  1. Red blood cell (RBC) folate concentrations.
  2. Total serum folate concentrations.
  3. The relative contribution of folate vitamers to total serum folate concentrations (unmetabolized folic acid, tetrahydrofolic acid, 5,10-methenylTHF, 5-formylTHF, 5-methylTHF and MeFox).
Time Frame: From FACT randomization at 8-16 weeks gestation to date of sample collection taken at one time point between 24 and 26 completed weeks gestation.
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | FACT High-dose Folic Acid Treatment Group | FACT Placebo Treatment Group
Number analyzed (Participants) | 19 | 31
nmol/L
  RBC folate | 2701 [2559 to 3017] | 2686 [2311 to 3047]
  Serum total folate by protein binding assay | 105 [57 to 183] | 67.1 [58.5 to 89]
  Serum total folate by LC-MS/MS | 148.4 [110.4 to 181.2] | 122.8 [99.5 to 136.0]
  5-MethylTHF | 126.6 [98.8 to 158.6] | 108.6 [96.4 to 123.2]
  unmetabolized folic acid | 4.6 [2.5 to 33.8] | 1.9 [0.9 to 4.1]
  THF | 3 [1 to 12.6] | 2.4 [0.6 to 8.5]
  5-formylTHF | 1.3 [0.8 to 1.6] | 1.4 [0.6 to 1.6]
  5,10-MethenylTHF | 0.9 [0.5 to 1.6] | 0.8 [0.2 to 1.0]
  MeFox | 6.9 [3.6 to 10.1] | 5.0 [2.4 to 8.0]

2. Secondary Outcome: Homocysteine Status
Description: Maternal homocysteine concentrations will be determined.
Time Frame: as for outcome 1
Population: Two participants in the High-dose Folic Acid Treatment Group and one participant in the Placebo Treatment Group had missing data for this outcome.
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | FACT High-dose Folic Acid Treatment Group | FACT Placebo Treatment Group
Number analyzed (Participants) | 17 | 30
nmol/L | 6 [4.6 to 7] | 6.4 [5.6 to 7.8]

3. Secondary Outcome: Status of Modifiers of Folate metabolism_vitamin B-12
Description: Status of modifiers of folate metabolism will be determined by Vitamin B6 and B12 concentrations
Time Frame: Taken at one time point between 24 and 26 completed weeks gestation.
Population: For Vitamin B-12 measurement, sample data are not available for one participant in the high-dose folic acid treatment group, and one participant in the placebo treatment group.
  Missing data are due to insufficient sample volume or compromised sample quality.
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | FACT High-dose Folic Acid Treatment Group | FACT Placebo Treatment Group
Number analyzed (Participants) | 18 | 30
pmol/L | 217.5 [191 to 271] | 208.5 [192 to 277]

4. Secondary Outcome: Angiogenic Potential
Description: Angiogenic potential will be determined from measurement of maternal circulating s-FLT-1, s-ENG-1 and placental growth factor concentrations.
Time Frame: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | FACT High-dose Folic Acid Treatment Group | FACT Placebo Treatment Group
Number analyzed (Participants) | 19 | 31
pg/mL
  Placenta growth factor (PlGF) | 421.4 [220.4 to 653.2] | 331.2 [214.2 to 580.7]
  soluble fms-like tyrosin kinase 1 (sFlt-1) | 862.9 [630.2 to 1382.2] | 812 [624.5 to 1381.0]
  soluble endoglin (sEng-1) | 961.5 [688.7 to 1250.1] | 1061.0 [669.9 to 1322.8]

5. Secondary Outcome: Status of Modifiers of Folate metabolism_MTHFR Genotype (C677T)
Description: Status of modifiers of folate metabolism will be determined by frequency of single nucleotide polymorphisms (SNPs) in the key folate metabolic enzyme MTHFR
Time Frame: Taken at one time point between 24 and 26 completed weeks gestation.
Population: The baseline distribution of MTHFR (C677T) genotype frequencies, ie, CC, TT, and CT are describe in each row.
Measure: Count of Participants; unit: Participants
Arm/Group | FACT High-dose Folic Acid Treatment Group | FACT Placebo Treatment Group
Number analyzed (Participants) | 19 | 31
Participants
  CC | 7 | 12
  CT | 9 | 15
  TT | 3 | 4

6. Secondary Outcome: Status of Modifiers of Folate metabolism_ Vitamin B6 (Pyridoxal 5-phosphate)
Description: Status of modifiers of folate metabolism will be determined by Vitamin B6 and B12 concentrations
Time Frame: Taken at one time point between 24 and 26 completed weeks gestation.
Population: For Vitamin B-6 (pyridoxal 5-phosphate), sample data are not available for one participant in the high-dose folic acid treatment group.
  Missing data are due to insufficient sample volume or compromised sample quality.
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | FACT High-dose Folic Acid Treatment Group | FACT Placebo Treatment Group
Number analyzed (Participants) | 18 | 31
nmol/L | 44.3 [19.0 to 71.4] | 40.0 [21.2 to 80.9]

ADVERSE EVENTS:
Arm/Group | FACT High-dose Folic Acid Treatment Group | FACT Placebo Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/31
Other Adverse Events (participants affected / at risk) | 0/19 | 0/31

LIMITATIONS AND CAVEATS:
Selection bias and generalizability: convenience sample from a larger trial of individuals at high risk for preeclampsia

Small sample size

Lack of baseline folate measurements and the single time-point evaluation of folate status: prevents analysis of changes in folate status and 1-carbon metabolism over the course of pregnancy

Samples were non-fasting and information on the timing of sample collection relative to ingestion of the daily folic acid supplements was not collected

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No